CLINICAL TRIAL: NCT03073993
Title: Nasogastric Versus Orogastric Route of Feeding in Preterm (<32 Weeks) Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Max Super Speciality Hospital (Other)
Responsible Party: Principal Investigator, SYED AHMAD ZIA, DNB Resident in Pediatrics, Max Super Speciality Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NGOG
Record Dates: First submitted 2016-08-02; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Apnea Prematurity
Keywords: nasogastric; orogastric; nutrition; preterm; feeding tube; insertion; episodes; bradycardia; desaturation
MeSH Terms: conditions — Premature Birth; Bradycardia | interventions — Intubation, Gastrointestinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasogastric (Active Comparator): Feeding tube insertion in nasogastric group
  Interventions: Procedure: feeding tube insertion
- Orogastric (Active Comparator): Feeding tube insertion in orogastric group
  Interventions: Procedure: feeding tube insertion

INTERVENTIONS:
Procedure: feeding tube insertion — Feeding tube was inserted in hemodynamically stable babies for purpose of feeding

SUMMARY:
Enteral feeding tubes in newborns are used for feeding preterm and low birth weight babies in neonatal intensive care units as they often do not suck effectively owing to lack of coordination between sucking, swallowing and breathing due to neurological immaturity and delayed gastric emptying.

The feeding tubes could be inserted by the nasogastric (NG) route or by the orogastric (OG) route. Both routes are used in different Neonatal Intensive Care Units (NICUs). Both methods are associated with different adverse events.

Since newborn infants are obligate nose breathers, nasogastric tube (NGT) can lead to partial nasal obstruction which might increase airway resistance and work of breathing although they are easy to secure to the face than orally placed tubes. Orogastric tubes (OGT), on the other hand, may not lead to the potential risk of increased work of breathing associated with NGT but are more frequently malpositioned and can loop inside the mouth. Also there is increased possibility of apnea and bradycardia due to vagal stimulation.

Despite so many years of continuing debate, the evidence of superiority of one method over another is not proven. Very few studies have tried to look into this matter and there are no consensus guidelines. This study is being conducted to compare the rate and type of adverse events in OG versus NG feeds in preterm neonates ≤ 32 weeks and postmenstrual age (PMA) ≤ 36 weeks.

Preterm neonates born at ≤ 32 weeks with PMA≤ 36 weeks who require feeding tube as a route for enteral feeding once they are out of respiratory support ( i.e ventilation or CPAP) are eligible candidates. Feeding tube insertion episode (FTIE) is defined as episode of insertion of OG or NG tube. FTIE will be randomized into NG or OG routes. Primary outcome is frequency of desaturation and bradycardia in each group.

DETAILED DESCRIPTION:
After written informed consent by either of the parent, preterm neonate (≤32 weeks gestational age and PMA ≤36weeks) fulfilling the inclusion criteria will be enrolled in the study if they require tube feeding.

Each episode of insertion of either NGT or OGT will be labelled as Feeding tube insertion episode (FTIE) in the study. Total of 160 FTIE will be done in study period, 80 FTIEs in preterm neonates of <30 weeks gestational age and 80 FTIE in preterm neonates of ≥30 weeks gestational age.

The method of FTIE (whether NG or OG) will be randomized into 2 groups by computer generated random sequence in blocks of 4 each. Stratification will be done as per Gestational age< 30 weeks and ≥ 30 weeks. Randomization sequence will be stored in sealed opaque envelope which was kept with one person who will not involved in care of patients.

Tube insertion will be done by NICU nursing staff who are already trained and validated in putting tube. Length of NGT/OGT insertion will be calculated by distance from bridge of nose to ear lobe and then from ear lobe to midway between xiphisternum and umbilicus (NEMU method). Correct tube placement will be checked by first aspirating and then pushing in 2 ml air and listening by stethoscope.

Each FTIE will be followed till the tube required to be changed for any reason, or tube feeding terminated due to graduation to direct feeds by paladay or breast. If the tube is changed for any reason, the reinsertion of the tube will be taken as a fresh FTIE, and again followed as above.

To record adverse events, heart rate and oxygen saturations will be recorded in the monitor till the time tube remained in situ. Bradycardia is defined as Heart rate < 100/min. Desaturation is defined as SpO2 < 85%. Alarms on the multifunction monitors (Philips MP 20 Neonatal) will be set with lower limit of Heart rate as 100/min and lower limit of saturation as 85%. Episodes will be recorded on a proforma lying at bedside by the duty nurse on the data collection form which include demographic parameters notably name, age, sex, IP No, gestational age at birth in weeks+ days, PMA at enrollment (weeks+ days), method of feeding (OG or NG) along with clinical parameters in the form of desaturation episodes/hr and bradycardia episodes/hr.

If a tube remained in situ for more than 24 hours, a new sheet will be taken. Each time monitor give alarm for desaturation and/ or bradycardia, nurse will check the baby and monitor. If the waveform showed regular trend and probe is attached properly to baby, episode will be recorded. Since the duration of NG and OG tubes may vary, the number of episodes of bradycardia and /or desaturation episodes/hr will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Hemodynamically stable preterm neonates (≤32 weeks gestational age and PMA ≤ 36weeks) not requiring respiratory support (CPAP/Heated humidified high flow oxygen/ Ventilation).

Exclusion Criteria:

* Babies (> 32 weeks and PMA>36 weeks)
* Severe congenital malformations, chromosomal abnormalities
* Baby requiring any respiratory support
* Sepsis, IVH, NEC or any illness explaining apneas

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Heart rate and saturation | 48 hours
  frequency of episodes of heart rate <100 and sauration < 85%

SECONDARY OUTCOMES:
infant feeding tube | 48 hours
  duration in hours after which it needs to be changed. We want to see whether nasogastric tube remains in situ for longer time or vice versa

CONTACTS AND LOCATIONS:
Overall Officials: Naveen P Gupta, MD, DNB, Study Director — Consultant Neonatologist

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bohnhorst B, Cech K, Peter C, Doerdelmann M. Oral versus nasal route for placing feeding tubes: no effect on hypoxemia and bradycardia in infants with apnea of prematurity. Neonatology. 2010;98(2):143-9. doi: 10.1159/000279617. Epub 2010 Mar 16. PMID 20234138